CLINICAL TRIAL: NCT00653484
Title: Energy Balance Interventions for Colorectal Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Maciej Buchowski, Research Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000592809; VU-VICC-GI-0810; VU-VICC-061020
Record Dates: First submitted 2008-04-04; First posted 2008-04-07 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer; Obesity
Keywords: colon cancer; rectal cancer; obesity
MeSH Terms: conditions — Colorectal Neoplasms; Obesity; Colonic Neoplasms; Rectal Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Physical Activity Only (Experimental): Physical Activity
  Interventions: Behavioral: Physical Activity
- Dietary Energy Restriction (Experimental): Energy restriction
  Interventions: Behavioral: Energy Restriction
- Physical Activity+Dietary Energy Restriction (Experimental): Physical Activity ad Energy Restriction
  Interventions: Behavioral: Physical Activity and Energy Restriction

INTERVENTIONS:
Behavioral: Physical Activity
  Arms: Physical Activity Only
Behavioral: Energy Restriction
  Arms: Dietary Energy Restriction
Behavioral: Physical Activity and Energy Restriction
  Arms: Physical Activity+Dietary Energy Restriction

SUMMARY:
RATIONALE: Calories and physical exercise may affect the risk of developing cancer. It is not yet known whether a low-calorie diet and/or physical activity program is effective in preventing cancer in participants at increased risk of developing colorectal cancer.

PURPOSE: This randomized clinical trial is studying diet and physical activity in healthy overweight, obese, or inactive participants at risk of developing colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare four 12-week energy-balance interventions comprising a physical activity intervention (+2,000 kcal/wk), a dietary energy restriction intervention (DER)(-2,000 kcal/wk), or a combined physical activity and DER intervention (+1,000/-1,000 kcal/wk) vs no intervention in healthy, overweight, or moderately obese participants at increased risk for developing colorectal cancer.
* To quantify changes in circulating biomarkers (e.g., insulin, IGF-1, leptin, c-reactive protein, or isoprostanes) proposed to mediate the anticarcinogenic effects of DER in these participants.

OUTLINE: This study consists of a 2-week run-in period (baseline) followed by a 12-week intervention period.

Participants undergo three study visits at Vanderbilt University General Clinical Research Center (GCRC). Beginning at study visit 1, participants undergo a 2-week run-in period to obtain baseline measures of body composition (via dual x-ray absorptiometry), cardiorespiratory fitness (via treadmill testing), physical activity, dietary intake, energy expenditure, and metabolic activity. Dietary assessments using 24-hour dietary recalls are conducted by the GCRC dietitian during the run-in period. GCRC dietitians complete three 24-hour recalls on randomly selected days during the 2-week assessment period to provide an estimate of the participant's habitual food intake at baseline. Baseline energy needs are assessed during activity monitored run-in period to obtain measures of the participant's resting energy expenditure and total daily energy expenditure. Participants are also assessed using a brief psychological profile that is used to individualize the study intervention for each participant.

Approximately 10-14 days after the initial visit and after all baseline assessments have been completed, participants undergo a second study visit. Participants are randomized to 1 of 4 intervention arms.

* Arm I (physical activity): Participants undergo an in-person, 30- to 60-minute counseling visit, followed by five brief 10- to 15-minute telephone-counseling calls over 12 weeks. During the initial counseling session, participants learn about goal setting and how to develop a personalized plan for meeting their intervention goals. Participants are instructed about wearing proper shoes and about monitoring their exercise duration and intensity. Participants are also given pedometers to help track their activity patterns and to monitor their progress in meeting program objectives. Participants must wear the pedometers for 7 days at baseline and again at 12 weeks. The information provided is used to estimate overall physical activity energy expenditure (PAEE), steps per day, and time spent in different levels of activity.

Participants are monitored periodically for adherence to the exercise program through behavioral counseling and self-reported logs of daily exercise and pedometer steps. Dietary intake is measured periodically using multiple 24-hour dietary recalls to carefully assess possible changes in energy intake and dietary quality over the course of the study.

* Arm II (dietary energy restriction [DER]): Based on the initial estimate of energy needs determined during the run-in period, participants receive a reduced-calorie, food exchange-based diet for 12 weeks. Each diet is individualized to achieve the desired daily energy deficit of 300 calories per day based on physical activity levels. All meals are prepared by the GCRC metabolic kitchen. Participants receive one multivitamin per day and no other nutritional supplements. Fluids including coffee, water, and other drinks are allowed at the pre-study level. Each week, participants meet with the dietitian to discuss the participant's progress, submit daily reports of food intake, return uneaten food items, and to provide urine samples for assessment of urinary biomarkers.

Adherence to the diet is monitored by compliance with food pick-up, dietary records, and measures of urinary metabolites. Participants are also provided with individual instruction, counseling, and assessment by the study dietitian.

* Arm III (physical activity and DER): Participants undergo a 12-week DER and physical-activity program, as described in arms I and II, with the exception that the dose of PAEE and DER in the combined intervention (i.e., +1,000/-1,000 kcal/week) is half that of each individual intervention (+2,000 kcal/week for arm I and -2,000 kcal/week for arm II). Participants in arm III receive an individualized reduced-calorie diet designed to achieve a desired daily energy deficit of 150 calories per day based on participant physical activity levels.
* Arm IV (wait-list control): Participants are followed periodically. At study visit 3, after completion of the 12-week study interventions, participants undergo repeat assessment of body composition, fitness, diet, and activity measures.

Participants undergo blood and urine sample collection at baseline and at 12 weeks for correlative laboratory studies. Blood samples are assessed for circulating biomarkers that are involved in energy homeostasis and metabolic control (e.g., insulin, IGF, and leptin) and inflammation and oxidative stress (e.g., c-reactive protein, PGE-2, and isoprostanes). Urine samples are examined for biomarkers of dietary protein intake (i.e., nitrogen content), dietary sodium, and potassium intake.

Participants complete the Community Health Activities Model Program for Seniors Physical Activity Questionnaire at baseline and at 12 weeks for assessment of PAEE through non-occupational activities, including social activities, recreation, hobbies, housework, walking, jogging, and 14 other types of exercise.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Healthy participants at increased risk for developing colorectal cancer due to any of the following risk factors:

  * Excess weight or obesity

    * Body mass index 25-40 kg/m²
  * Not currently exercising on a regular basis (< 1,000 kcal/week)
* Must be free of significant eating disorders (i.e., purging, extended fasting, or use of laxatives)

PATIENT CHARACTERISTICS:

* Females must be postmenopausal, defined by the absence of menstrual periods in the past 12 months
* No heart disease or orthopedic impairments that would limit exercise or may be worsened by exercise
* No major chronic diseases (e.g., liver, kidney, diabetes, or adrenal ailments) that would influence metabolism
* No cancer diagnoses within the past 5 years, except skin cancer

Exclusion Criteria:

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Physical activity-energy expenditure | June 2010

SECONDARY OUTCOMES:
Physical activity-energy expenditure | June 2010
Dietary-energy intake (kcal/d) and quality | June 2010
Body weight and composition | June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Charles Matthews, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee